CLINICAL TRIAL: NCT02368288
Title: Efficacies of Entecavir Add on Chronic Hepatitis B Patients With HBV DNA Load ≥1000 Copies/ml After 6 Months Treatment of Peginterferon Alpha 2a
Brief Title: Efficacies of Entecavir Add on HBeAg Positive Patients With HBV DNA Positive During Peginterferon Alpha 2a Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, liver disease center, Beijing Ditan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DTXY005
Record Dates: First submitted 2015-02-14; First posted 2015-02-23 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Hepatitis B
Keywords: chronic hepatitic B; peginterferon; HBsAg; entecavir
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- entecavir with PEG-IFN a-2a (Experimental): after enrolled, entecavir will added, and patients will receive treatment of PEG-IFN a-2a combine with entecavir for 48 weeks.
  Interventions: Drug: entecavir
- peginterferon alpha 2a (No Intervention): in this group, patients will be continue treated only with PEG-IFN a-2a for 48 weeks after enrolled.

INTERVENTIONS:
Drug: entecavir — in this group, entecavir will added, and patients will receive treatment of PEG-IFN a-2a combine with entecavir for 48 week.
  Arms: entecavir with PEG-IFN a-2a

SUMMARY:
The aim of interferon therapy in HBeAg positive chronic hepatitis B was to make patients obtain immune control to hepatitis B virus defined as occurred HBeAg seroconversion and HBsAg loss with sustained viral response after treatment. However this target could not be get if patients keep HBV DNA positive during interferon treatment and offend relapse after withdraw of treatment. In this trail, Nucleoside(acid) analogues(NA) will add on patients with HBV DNA load ≥1000copies/ml after 6 months of interferon treatment, and the efficacies of the combine therapy were evaluated by the rates of HBeAg seroconversion and HBsAg loss after 48 weeks of combined therapy, compared with control group.

DETAILED DESCRIPTION:
HBeAg positive patients with HBV DNA load ≥1000copies/ml after 6 months of peginterferon alpha 2a treatment will be enrolled randomized into two groups, in intervention group, patients will receive entecavir combine with peginterferon alpha 2a(PEG-IFN a-2a) treatment for 48 weeks and follow 24 weeks. Patients in control group will be continue treated with PEG-IFN a-2a for 48 weeks and followed 24 weeks. Serum HBV DNA load, HBsAg/anti-HBs level, HBeAg/anti-HBe will be tested at enrollment and every 3 months during the treatment course. Parameters of Liver and kidney function, and liver ultrasound examination will be tested with intervals 1-3 months. The efficacies of the combined therapy were evaluated by the rates of HBeAg seroconversion and HBsAg loss after 48 weeks of combined therapy, compared with control group.

ELIGIBILITY:
Inclusion Criteria:

* HBeAg positive patients with HBV DNA load ≥1000copies/ml after 6 months of peginterferon a-2a treatment

Exclusion Criteria:

* Active consumption of alcohol and/or drugs
* Co-infection with human immunodeficiency virus, hepatitis C virus, or hepatitis D virus
* History of autoimmune hepatitis
* Psychiatric disease
* Evidence of neoplastic diseases of the liver

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
rate of HBeAg seroconversion | 48 weeks
  HBeAg seroconversion defined as HBeAg loss with anti-HBe antibody positive was evaluated during weeks treatment period

SECONDARY OUTCOMES:
rate of HBsAg loss | 48 weeks
  HBsAg loss defined as HBsAg level ≤0.05 IU/ml after 48 week treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan hospital,Capital Medical University, Beijing, Beijing Municipality, China